CLINICAL TRIAL: NCT06171685
Title: A Phase II Randomized Adaptive Platform Trial Evaluating Novel Therapies in Relapsed or Refractory Multiple Myeloma
Brief Title: MMRC Horizon One Adaptive Platform Trial Evaluating Therapies in RRMM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Multiple Myeloma Research Consortium (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MMRC-099
Record Dates: First submitted 2023-11-03; First posted 2023-12-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-01

CONDITIONS: Relapse Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sub-protocol A (Active Comparator): Serves as the reference arm for the platform
  Interventions: Drug: Teclistamab Monotherapy
- Sub-Protocol B (Experimental): This arm will be an investigational arm
  Interventions: Drug: Teclistamab

INTERVENTIONS:
Drug: Teclistamab Monotherapy — standard of care
  Other Names: Tecvayli
  Arms: Sub-protocol A
Drug: Teclistamab — investigational doses compared to SOC
  Other Names: Tecvayli
  Arms: Sub-Protocol B

SUMMARY:
This trial is an adaptive platform trial. The structure of the protocol allows the trial to evolve over time. Multiple investigational arms will be included within the trial under a Master Protocol (MP). These investigational arms may be added as appendices at different times depending on whether they are trial-ready and whether accrual in the trial will support another arm. Accrual to an arm will terminate in accord with the arm's appendix to the Master Protocol.

The purpose of this proposed structure is to support the recurrent research challenge of efficiently evaluating what is the best therapy for a particular patient.

ELIGIBILITY:
Inclusion Criteria

For inclusion in the trial, all the following inclusion criteria must be fulfilled, as no waivers will be permitted:

* Voluntarily agree to participate by giving written informed consent
* ≥18 years of age
* Histologically confirmed multiple myeloma that is exposed, relapsed, or intolerant to one of each of the following classes of agents:

  * A proteasome inhibitor
  * An immunomodulatory drug
  * An anti-CD38-monoclonal antibody
  * Must have received between 1-4 lines of prior systemic therapy
  * Prior BCMA-directed antibody-drug conjugate (ADC) or chimeric antigen receptor (CAR)-T cell therapy allowed Note: A washout period of 6 months is required from prior anti-BCMA therapy. For BCMA CAR-T cell therapy, participants must be ≥ 6 months from lymphodepleting chemotherapy.
* Measurable disease, defined as one of the following:

  * M-protein ≥ 0.50g/dL (0.5 g/dL or above if IgA subtype)
  * Urine M-protein (Bence-Jones protein) ≥ 200 mg/24hours
  * Serum free light chain difference > 100 mg/L
  * Biopsy proven plasmacytoma
* For oligosecretory multiple myeloma, disease must be measurable by imaging (i.e., PET-CT, MRI)
* ECOG performance status of 0-2
* Adequate organ function, as indicated by the following laboratory values:

  * Adequate hematological function, defined as ANC ≥ 1000/µL, platelet count ≥ 50,000/µL, and hemoglobin ≥ 8 g/dL (transfusion and/or growth factor support is allowed for hematologic parameters as long as the investigator deems the participant otherwise fit for screening)
  * Adequate hepatic function, defined as total bilirubin level < 1.5 x institutional upper limit of normal (IULN) (except in participants with congenital bilirubinemia, such as Gilbert syndrome, in which case direct bilirubin < 1.5-3.0 x IULN is required), AST ≤ 2.5 x IULN, and ALT ≤ 2.5 x IULN
  * Adequate renal function, defined as calculated creatinine clearance ≥ 30 mL/min per institutional standard (assessment method should be recorded, measured or C-G acceptable)
  * eGFR > 30mL/min based on MDRD 4-variable formula calculation or creatinine clearance based measured by 24h urine collection
  * Corrected serum calcium <14mg/dL or free ionized calcium <6.5 mg/dL
* Persons of childbearing potential must have a negative serum pregnancy test at screening (within 72 hours of first dose of trial medication). Non-childbearing potential for a person assigned as female at birth is defined as 1 of the following:

  * ≥ 45 years of age and has not had menses for >1 year
  * Amenorrheic for > 2 years without a hysterectomy and/or oophorectomy and follicle-stimulating hormone value in the postmenopausal range upon pretrial (screening) evaluation
  * Status is post-hysterectomy, -oophorectomy, or -tubal ligation
* Persons of childbearing potential must be willing to use highly effective contraceptive measures during sexual contact with a person assigned as male at birth starting with the Screening visit through 90 days after last dose of trial medication.

Note: Abstinence is acceptable if this is the established and preferred contraception for the participant.

-Persons assigned as male at birth with a partner(s) of childbearing potential must agree to use highly effective contraceptive measures throughout the trial starting with the Screening visit through 90 days after the last dose of trial medication is received. Persons assigned as male at birth with pregnant partners must agree to use a condom; no additional method of contraception is required for the pregnant partner.

Note: Abstinence is acceptable if this is the established and preferred contraception method for the participant.

* Known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using New York Heart Association Functional Classification. To be eligible for this trial, participants should be Class 2 or better. Class 2 is defined as slight limitation of physical activity, in which ordinary physical activity leads to fatigue, palpitation, or dyspnea; the person is comfortable at rest.
* Prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessments of the investigational arms are eligible for this trial.
* Known HIV infection who are on effective anti-retroviral therapy with undetectable viral load within 6 months of screening and enrollment are eligible for this trial.
* Evidence of chronic hepatitis B virus (HBV) infection must have an undetectable HBV viral load on suppressive therapy, if indicated.
* History of hepatitis C virus (HCV) infection must have been treated and cured. For participants with known HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Willing and able to comply with the requirements of the protocol.

Exclusion Criteria

For inclusion in Horizon, participants will not be eligible if any of the following criteria are met, as no waivers will be permitted:

* Major concurrent illness or organ dysfunction including but not limited to the following:

  * Plasma cell leukemia (the presence of ≥ 5% circulating plasma cells in peripheral blood smears)
  * Waldenström's macroglobulinemia
  * POEMS syndrome
  * Primary amyloid light-chain amyloidosis
* History of allergy or known hypersensitivity to any of the trial therapies or any of their excipients, or contraindication to any of the trial therapies as outlined in the local prescribing information (e.g., United States Prescribing Information [USPI]).
* Complete cord compression or CNS involvement
* Active or history of autoimmune disease that requires systemic treatment within 2 years of the start of study drug (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs).

Note: Participants with diabetes type 1, vitiligo, psoriasis, or hypo- or hyperthyroid disease not requiring immunosuppressive treatment are eligible

* Received a live, attenuated vaccine within 4 weeks before the first dose of study drug. Non-live or nonreplicating vaccines authorized for emergency use (eg, COVID-19) by local health authorities are allowed.
* Allogeneic tissue/solid organ transplant recipients with chronic GVHD requiring steroid equivalent dose of > 20 mg prednisone
* Active infection requiring treatment
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the trial
* Legally incapacitated or has limited legal capacity
* Persons who are pregnant or lactating

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-11-17 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
ORR | through completion of the study, and yearly
  Objective Response Rate

CONTACTS AND LOCATIONS:
Overall Officials: Hearn J Cho, MD, PhD, Principal Investigator — Multiple Myeloma Research Foundation
Locations (13):
- United States (13):
  - City of Hope, Duarte, California
  - Emory Winship Cancer Center, Atlanta, Georgia
  - University of Chicago Cancer Center, Chicago, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute/Harvard Medical School, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Center, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Mt. Sinai School of Medicine, New York, New York
  - Atrium Levine Cancer Institute, Charlotte, North Carolina
  - Tennessee Oncology, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No